CLINICAL TRIAL: NCT01570868
Title: Ponatinib as Initial Therapy for Patients With Chronic Myeloid Leukemia in Accelerated Phase
Brief Title: Ponatinib - Frontline for Chronic Myeloid Leukemia (CML) in Accelerated Phase (AP)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0074; NCI-2012-00572 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-02

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic Myeloid Leukemia; CML; Chronic Phase; Cytogenetic response; CCyR; Major molecular response; MMR; Complete molecular response; CMR; Ponatinib; AP24534
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Intervention Model Description: Participants enrolled before July 25, 2013 were given a starting dose of 45 mg per day. The study was amended and the dose was lowered due to tolerability. Participants enrolled after this date were given a starting dose of 30 mg per day.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ponatinib 45 mg (Experimental): Ponatinib at a dose of 45 mg orally, once daily. If a dose is missed or vomited, the next dose should not be increased to account for missing a dose. Total duration of therapy 3 to 5 years.
  Interventions: Drug: Ponatinib
- Ponatinib 30 mg (Experimental): Ponatinib at a dose of 30 mg orally, once daily. If a dose is missed or vomited, the next dose should not be increased to account for missing a dose. Total duration of therapy 3 to 5 years.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Starting dose: 45 mg by mouth once daily.
  Other Names: AP24534

SUMMARY:
The goal of this clinical research study is to learn if ponatinib can help to control Chronic Myeloid Leukemia (CML) in accelerated phase. The safety of this drug will also be studied.

Ponatinib is designed to block the function of BCR-ABL, which is the abnormal protein responsible for causing leukemia in certain cells.

Ponatinib may cause a blood clot to form in an artery or in a vein. Depending on the location of the clot, this could cause a heart attack, a stroke, severe damage to other tissue, or death. A blood clot may occur within 2 weeks after you start taking the drug. About 25% (1 in 4) of patients taking the drug form an abnormal clot. Blood clots can occur in patients that do not have other known risk factors for forming clots. If you develop a blood clot, you will need to stop taking ponatinib. In some cases, emergency surgery could be needed to remove the clot and restore blood flow.

DETAILED DESCRIPTION:
Study Drug Administration:

You will take ponatinib by mouth 1 time every day while you are on study with about a cup (8 ounces) of water. You should not eat within 2 hours before or after taking the drug. You will complete a study diary in which you will record the date and time that you take the study drug each time. If you miss any doses, you will also note this in the study diary. Bring this diary to every study visit, as described below.

Study Visits:

The tests and procedures for this study have a wide range of time in which they can be done. In general, your schedule of study visits will be as follows:

* Weekly in Month 1
* Monthly in Year 1
* Three (3) to 4 times in Year 2
* Two (2) to 3 times in every year after that

The study staff will help you schedule your study visits. The following tests and procedures will be performed:

* Every 1-2 weeks for the first 4 weeks, then every 4-6 weeks for the first year, then every 3-4 months for the next year, then every 4-6 months after that, blood (about 1/2 tablespoon) will be drawn for routine tests.
* Every 3 months for the first year, you will have an ECG.
* Every 3 months for the first year, then every 6-12 months after that, you will have a physical exam.
* Every 3-4 months for the first year, then every 6-12 months after that, blood (about 2 teaspoons) will be drawn to measure levels of leukemia cells in your body.
* Every 3-4 months for the first year, then every 6-12 months for the next 2 years, then every 2-3 years after that, you will have a bone marrow aspirate for genetic testing and to check the status of the disease.

Length of Participation:

You may continue taking the study drug for up to 5 years. You will be taken off study early if intolerable side effects occur, if the disease gets worse, or if you are unable to follow study directions.

Your participation on the study will be over when you have completed the follow-up visit/call.

Follow-Up:

If you leave the study, you will be called or you will come to the clinic within 30 days to learn about any side effects or symptoms you may be having. If you are called, this call will last about 2-3 minutes.

This is an investigational study. Ponatinib is FDA approved to treat patients with certain types of leukemia. Its use in this study is investigational.

Up to 80 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Ph-positive (by cytogenetics or FISH) or Bcr-ABL-positive (by PCR) CML with accelerated phase features at the time of diagnosis.
2. Patients must have received no or minimal prior therapy, defined as </=1 month of prior IFN-α (with or without ara-C) and/or an FDA-approved tyrosine kinase inhibitor (e.g, dasatinib, nilotinib). Prior use of hydroxyurea or anagrelide is allowed with no limitations.
3. Age >/=18 years
4. Eastern Cooperative Oncology Group (ECOG) performance of 0-2.
5. Adequate end organ function, defined as the following: total bilirubin <1.5x upper limit of normal (ULN), serum glutamate pyruvate transaminase (SGPT) <2.5x ULN,creatinine clearance (CrCl) >/= 30 mL/min at screening (calculation according to Cockcroft & Gault formula).
6. Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
7. Women of pregnancy potential must practice an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control. Adequate forms of contraception are barrier methods (e.g., condoms, diaphragm), oral, depo provera, or injectable contraceptives, intrauterine devices, spermicidal jelly or foam, abstinence, and tubal ligation. Women and men must continue birth control for the duration of the trial & at least 3 months after the last dose of study drug.
8. **continued from above: All WOCBP MUST have a negative serum or urine pregnancy test within 7 days prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.

Exclusion Criteria:

1. NYHA cardiac class 3-4 heart disease
2. Cardiac Symptoms: Patients meeting the following criteria are not eligible: History of unstable angina, myocardial infarction, transient ischemic attack (TIA), stroke, peripheral arterial occlusive disease, venous thromboembolism or pulmonary embolism; Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes); Prolonged corrected QT interval (QTc) interval on pre-entry electrocardiogram (> 470 msec) on both the Fridericia and Bazett's correction; Symptomatic congestive heart failure within 3 months prior to first dose of ponatinib (NYHA class III or IV).
3. Patients with active, uncontrolled psychiatric disorders including: psychosis, major depression, and bipolar disorders.
4. Pregnant or breast-feeding women are excluded.
5. Patients with uncontrolled hypertension (defined as sustained stage 2 hypertension, i.e., systolic BP >/=160 mmHg or diastolic BP >/=100 mmHg).
6. Patients with history of pancreatitis.
7. Patients in late chronic phase (i.e., time from diagnosis to treatment >6 months), or blast phase are excluded. The definitions of CML phases are as follows: A. Early chronic phase: time from diagnosis to therapy </= 6 months; B. Late chronic phase: time from diagnosis to therapy > 6 months; C. Blastic phase: presence of 30% blasts or more in the peripheral blood or bone marrow; D. Accelerated phase CML: presence of any of the following features: Peripheral or marrow blasts 15% or more; Peripheral or marrow basophils 20% or more; Thrombocytopenia < 100 x 10(9)/L unrelated to therapy; Documented extramedullary blastic disease outside liver or spleen.
8. **continued from above: E. Clonal evolution defined as the presence of additional chromosomal abnormalities other than the Ph chromosome has been historically been included as a criterion for accelerated phase. However, patients with clonal evolution as the only criterion of accelerated phase have a significantly better prognosis, and when present at diagnosis may not impact the prognosis at all. Thus, patients with clonal evolution and no other criteria for accelerated phase will be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Kantarjian H, Boddu PC, Nogueras-Gonzalez GM, Verstovsek S, Garcia-Manero G, Borthakur G, Sasaki K, Kadia TM, Sam P, Ahaneku H, O'Brien S, Estrov Z, Ravandi F, Jabbour E, Cortes JE. Analysis of cardiovascular and arteriothrombotic adverse events in chronic-phase CML patients after frontline TKIs. Blood Adv. 2019 Mar 26;3(6):851-861. doi: 10.1182/bloodadvances.2018025874. PMID 30885996
- [Derived] Issa GC, Kantarjian HM, Gonzalez GN, Borthakur G, Tang G, Wierda W, Sasaki K, Short NJ, Ravandi F, Kadia T, Patel K, Luthra R, Ferrajoli A, Garcia-Manero G, Rios MB, Dellasala S, Jabbour E, Cortes JE. Clonal chromosomal abnormalities appearing in Philadelphia chromosome-negative metaphases during CML treatment. Blood. 2017 Nov 9;130(19):2084-2091. doi: 10.1182/blood-2017-07-792143. Epub 2017 Aug 23. PMID 28835440
- [Derived] Jain P, Kantarjian H, Jabbour E, Gonzalez GN, Borthakur G, Pemmaraju N, Daver N, Gachimova E, Ferrajoli A, Kornblau S, Ravandi F, O'Brien S, Cortes J. Ponatinib as first-line treatment for patients with chronic myeloid leukaemia in chronic phase: a phase 2 study. Lancet Haematol. 2015 Sep;2(9):e376-83. doi: 10.1016/S2352-3026(15)00127-1. PMID 26436130
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: April 27, 2012 to May 12, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early.
Groups:
- Ponatinib 45 mg: Ponatinib 45 mg orally, once daily.
- Ponatinib 30 mg: Ponatinib 30 mg orally, once daily.
Period: Overall Study
Arm/Group | Ponatinib 45 mg | Ponatinib 30 mg
Started | 43 | 8
Completed | 0 | 0
Not Completed | 43 | 8
Not completed — Adverse Event | 8 | 1
Not completed — FDA Recommendation | 23 | 3
Not completed — Physician Decision | 10 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponatinib 45 mg | Ponatinib 30 mg | Total
Number analyzed (Participants) | 43 | 8 | 51
Age, Continuous [Median (Full Range); unit: years] | 52 [21 to 74] | 42 [31 to 65] | 43 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 5 | 24
  Male | 24 | 3 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 8 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Cytogenetic Response (CCyR)
Description: Proportion of participants with previously-untreated accelerated phase CML attaining complete cytogenetic response (CCyR) at 6 months of treatment with Ponatinib classified according to suppression of the Philadelphia chromosome (Ph) by cytogenetics (FISH if cytogenetic analysis not informative, e.g., insufficient metaphases). CCyR defined as Ph positive 0%.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Ponatinib 45 mg: Ponatinib 45 mg orally, once daily. Dose escalation to 30 mg possible for participants with adverse events.
- Ponatinib 30 mg: Ponatinib 30mg orally, once daily. Dose escalation to 30 mg possible for participants with adverse events.
Arm/Group | Ponatinib 45 mg | Ponatinib 30 mg
Number analyzed (Participants) | 42 | 8
Participants | 40 | 3

2. Primary Outcome: Number of Participants With Complete Cytogenetic Response (CCyR)
Description: Proportion of participants with previously-untreated accelerated phase CML receiving treatment of Ponatinib achieving a Complete cytogenetic response (CCyR). Classified according to suppression of the Philadelphia chromosome (Ph) by cytogenetics (FISH if cytogenetic analysis not informative, e.g., insufficient metaphases. CCyR is defined as Ph positive 0%.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib 45 mg | Ponatinib 30 mg
Number analyzed (Participants) | 42 | 8
Participants | 42 | 6

3. Secondary Outcome: Toxicity Profile: Most Common Grade 3-4 Non-Hematologic Adverse Events (AEs) Seen in More Than 1 Participant
Description: Time to toxicity monitoring defined as any grade 3 or 4 drug-related non-hematologic adverse event that has not resolved to grade 2 or less after 6 weeks of optimal therapeutic management, or drug-related toxicity of any grade that in the opinion of the investigator prevents further therapy with ponatinib. Time to toxicity monitored using the Bayesian method of Thall, et al.
Time Frame: 3 months
Population: One participant was not included in analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Ponatinib 45 mg: Ponatinib oral dose 45 mg daily.
- Ponatinib 30 mg: Ponatinib oral dose 30 mg daily.
Arm/Group | Ponatinib 45 mg | Ponatinib 30 mg
Number analyzed (Participants) | 43 | 8
Participants
  Elevated Amylase | 2 | 0
  Lipase Elevation | 15 | 1
  Pancreatitis | 7 | 2
  Abdominal Pain | 1 | 0
  Hypertension | 3 | 0
  Elevated alanine aminotransferase (ALT) | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection minimally every 4 weeks for total duration of therapy up to one year, study collection period to be 3 to 5 years.
Arm/Group | Ponatinib 45 mg | Ponatinib 30 mg
Serious Adverse Events (participants affected / at risk) | 17/43 | 3/8
Other Adverse Events (participants affected / at risk) | 35/43 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib 45 mg (N=43) | Ponatinib 30 mg (N=8)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infections and infestations-Other (Infections and infestations) | 2 (2) | 0 (0)
Lung Infection (Infections and infestations) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Non-Cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 7 (10) | 2 (2)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Hysterectomy (Infections and infestations) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vaso-Occulusive diasease (Vascular disorders) | 1 (1) | 0 (0)
Bialteral superfical femoral artery occulsion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib 45 mg (N=43) | Ponatinib 30 mg (N=8)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac Disorders other (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased libido (Psychiatric disorders) | 1 (1) | 0 (0)
decreased range of motion, joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Increased Alanine aminotransferase (Investigations) | 2 (2) | 0 (0)
Increased amylase (Investigations) | 2 (2) | 0 (0)
Increased Aspartate aminotransferase (Investigations) | 1 (2) | 0 (0)
Increased GGT (Investigations) | 1 (1) | 0 (0)
Increased Lipase (Investigations) | 10 (15) | 1 (1)
Infection other (Infections and infestations) | 2 (2) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 7 (7) | 2 (2)
Pelvic infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 5 (5) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vascular disorders (Vascular disorders) | 3 (3) | 0 (0)
Weight gain (Investigations) | 3 (3) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes